CLINICAL TRIAL: NCT02177942
Title: A Double Blind Randomised Controlled Trial in Pre-school Age Children to Evaluate the Impact of a Nutritional Beverage Powder on Cognitive Performance Measures
Brief Title: A Clinical Trial to Study the Impact of a Nutritional Beverage on Tests of Memory in Healthy Preschool Age Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 202155; RH01722 (Other: GSK)
Record Dates: First submitted 2014-06-26; First posted 2014-06-30 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Cognition
MeSH Terms: interventions — Diet, Protein-Restricted

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test beverage powder (Experimental): 30 grams of cereal beverage powder with protein and added micronutrients will be made up to 100 mL drink using luke warm water. Subjects will be administered two doses of the drink (100 mL each) everyday
  Interventions: Other: Test beverage powder (High Proteins and added micronutrients)
- Control beverage powder (Active Comparator): 30 grams of cereal beverage powder with low protein and no added micronutrients will be made up to 100 mL using luke warm water. Subjects will be administered two doses of the drink (100 mL each) everyday
  Interventions: Other: Control beverage powder (Low protein and no added micronutrients)

INTERVENTIONS:
Other: Test beverage powder (High Proteins and added micronutrients) — High protein and added Micronutrients at recommended dietary allowance levels
  Arms: Test beverage powder
Other: Control beverage powder (Low protein and no added micronutrients) — Low protein and no added micronutrients
  Arms: Control beverage powder

SUMMARY:
The effect of supplementation using both protein and multiple micronutrients in preschool age children on cognitive performance and growth is unknown. The study will compare the effect of combination of protein and multiple micronutrients on indicators of cognitive performance and growth in preschool age children. Cognitive performance and anthropometric assessments will be measured at baseline and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Consent: Demonstrates understanding of the study and willingness to participate as evidenced by subject's parents or legally authorised representative's voluntary written informed consent and has received a signed and dated copy of the informed consent form.
2. Compliance : Understands and is willing, able and likely to comply with all study procedures and restrictions
3. General Health : Good general and mental health with, in the opinion of the investigator
4. Child with BMI for age between <+1 standard deviation (SD) to > -2SD

Exclusion Criteria:

1. Children in Care (CiC): A child who has been placed under the control or protection of an agency, organisation, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation.
2. Allergy/Intolerance: Known or suspected intolerance or hypersensitivity to the study materials (lactose, wheat gluten, soy protein) or any of their stated ingredients.
3. Child with severe anaemia (Haemoglobin < 7 g/dl) as determined by the non invasive spectrophotometry results.
4. Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit.
5. Participation in any nutritional study or didactic nutrition education in the last 6 months of the screening visit

5. Current or relevant history of any serious, severe or unstable physical or psychiatric illness or any medical disorder that would make the subject unlikely to fully complete the study or any condition that presents undue risk from the study product or procedures in the opinion of the investigator.

6. Recent history (3 months) of serious infections, injuries and/ or surgeries. 7. Children consuming iron, calcium and/or other nutritional supplements and/ or health food drinks on a regular basis (more than 3 times a week, in the recommended dosage) in the last 1 month prior to screening visit.

8. Use of any prescription medications during the study period for more than or equal to two weeks.

Ages: 36 Months to 65 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 528 (Actual)
Dates: Start 2014-06-20 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Karamsad, Gujarat, India

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at one center in India.
Pre-assignment Details: A total of 656 participants were screened out of which 528 were randomized to study treatments. 363 participants completed the study. Of the 165 randomized participants not completing the study, 152 withdrew consent, 10 participants violated the protocol, 2 participants were lost to follow up and 1 withdrew due to adverse event.
Groups:
- Test: 30 grams of cereal beverage powder with protein and added micronutrients was made up to 100 mililiters (mL) drink using luke warm water. Participants were administered two doses of the drink (100 mL each) everyday.
- Control: 30 grams of cereal beverage powder with low protein and no added micronutrients was made up to 100 mL using luke warm water. Participants were administered two doses of the drink (100 mL each) everyday.
Period: Overall Study
Arm/Group | Test | Control
Started | 262 | 266
Completed | 185 | 178
Not Completed | 77 | 88
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 4 | 6
Not completed — Withdrawal by Subject | 71 | 81

BASELINE CHARACTERISTICS:
Population: ITT population included all randomized participants who were administered at least one study treatment during the study and provided at least one post-baseline assessment of efficacy which was same as end of study (at 6 months). This analysis was conducted on ITT population. ITT (N=363)
Groups:
- Test: 30 grams of cereal beverage powder with protein and added micronutrients was made up to 100 mL drink using luke warm water. Participants were administered two doses of the drink (100 mL each) everyday.
- Total: Total of all reporting groups
Arm/Group | Test | Control | Total
Number analyzed (Participants) | 185 | 178 | 363
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.21 (0.607) | 4.24 (0.646) | 4.22 (0.626)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 66 | 149
  Male | 102 | 112 | 214

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Short Term Memory at 6 Months
Description: Short term memory was measured using word order and number recall sub tests of Kaufman Assessment Battery for Children (KABC).In Number Recall, child was asked to repeat series of number in same sequence after making sure that child is paying attention.A score of 0 and 1 given for incorrect and correct response respectively. In Word Order,qualified site staff said series of words and child then pointed pictures of those words in same sequence.Later items (object cards with pictures) included an interference task in which child named colors after hearing the word. Each subtest score was the total of item scores, ranging from 0-31 for word order and 0-22 for number recall. The two subtest scores were standardized for each subject and visit (Z score), and short term memory was calculated as the average of the two standardized values where higher scores reflect better short term memory.
Time Frame: Baseline and 6 months
Population: ITT population included all randomized participants who were administered at least one study treatment during the study and provided at least one post-baseline assessment of efficacy which was same as end of study (at 6 months). This analysis was conducted on ITT population.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Control: 30 grams of cereal beverage powder with low protein and no added micronutrients was made up to 100 mL drink using luke warm water. Participants were administered two doses of the drink (100 mL each) everyday.
Arm/Group | Test | Control
Number analyzed (Participants) | 185 | 178
Score on a scale | -0.04 (0.926) | -0.01 (0.856)
Statistical Analysis 1: Comparison: Test vs Control; Test type: Superiority or Other; p = 0.6931, ANCOVA; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.20 to 0.13] — Difference is test treatment minus control treatment such that a positive difference favours the test treatment

2. Secondary Outcome: Change From Baseline in Weight at 6 Months
Description: Weight was measured (single measurement) in standard clothing on weighing scale to the nearest 0.1kilograms(kg).
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Test | Control
Number analyzed (Participants) | 185 | 178
kg | 0.15 (0.436) | 0.14 (0.454)

3. Secondary Outcome: Change From Baseline in Height at 6 Months
Description: Height was measured (single measurement) using a portable stadio-meter, with the participant standing bare-foot, to the nearest 0.1centimeters (cm).
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Test | Control
Number analyzed (Participants) | 185 | 178
cm | 0.23 (0.442) | 0.20 (0.368)

4. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at 6 Months
Description: BMI for was obtained using the World Health Organization Anthroplus software version 1.0.2.
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Test | Control
Number analyzed (Participants) | 185 | 178
kg/m^2 | 0.00 (0.584) | 0.02 (0.634)

5. Secondary Outcome: Change From Baseline in Triceps Skin Fold (TSF) at 6 Months
Description: The TSF was measured in the midline of the posterior aspect of the arm, over the triceps muscle, at a level midway between the lateral projection of the acromion process of the scapula and the inferior margin of the olecranon process of the ulna. The right elbow is flexed at 90°and the midpoint between the acromion and the olecranon process is located and marked at the lateral side of the arm. The skinfold was then measured with the arm hanging loosely while standing. The triceps skinfold was picked up with the left thumb and index finger approximately 1cm proximal to the marked level and the tips calipers were applied to the skin-fold at the marked level. The triceps measurement was done (three measurements) using Holtain calipers to the nearest 0.2 millimeters (mm) and the average value was recorded.
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Test | Control
Number analyzed (Participants) | 185 | 178
mm | -0.33 (1.810) | -0.33 (2.062)

6. Secondary Outcome: Change From Baseline in Mid Upper Arm Circumference (MUAC) at 6 Months
Description: The MUAC (single measurement) was measured midway between the acromion and the olecranon process, while the participant stands with the elbow flexed at 90. The circumference was measured with a fiber glass tape to the nearest 0.1 cm on the right hand.
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Test Beverage Powder: 30 grams of cereal beverage powder with protein and added micronutrients was made up to 100 mL drink using luke warm water. Participants were administered two doses of the drink (100 mL each) everyday.
- Control Beverage Powder: 30 grams of cereal beverage powder with low protein and no added micronutrients was made up to 100 mL drink using luke warm water. Participants were administered two doses of the drink (100 mL each) everyday.
Arm/Group | Test Beverage Powder | Control Beverage Powder
Number analyzed (Participants) | 185 | 178
cm | 0.55 (1.131) | 0.57 (1.016)

7. Secondary Outcome: Change From Baseline in Arm Muscle Area (AMA) and Arm Fat Area (AFA) at 6 Months
Description: Using the MUAC measurement and TSF measurement, the arm muscle AMA and AFA were calculated i.e. AMA (cm2) = (MUAC-(π*TSF))2/4 π and AFA (cm2) = (MUAC2/4π) - AMA
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Centimeter square Cm^2
Arm/Group | Test | Control
Number analyzed (Participants) | 185 | 178
Centimeter square Cm^2
  Change from Baseline at 6 months (AMA) | 1.34 (2.770) | 1.39 (2.509)
  Change from Baseline at 6 months (AFA) | -0.01 (1.146) | 0.00 (1.330)

8. Secondary Outcome: Number of Ill Days at 6 Months
Description: Number of ill days due to cold, cough and/or associated fever were recorded. The mean number of ill days due was analyzed at 6 months using Analysis of Variance (ANOVA).
Time Frame: Baseline upto 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | Test | Control
Number analyzed (Participants) | 185 | 178
Number of days | 5.94 (3.130) | 7.45 (8.976)

9. Secondary Outcome: Change From Baseline in Problem Solving at 6 Months
Description: Test measured visual construction ability, understanding of spatial relationships and problem solving abilities. The child arranged flat shapes of various sizes and colors (items) to match a model or picture as instructed by the qualified staff. For items 1 to 2 (score 2 for success on first trial and 1 on second trial); items 3 to 10 (Score 1 for success and 0 for failure on first trial). The test continued till 3 consecutive scores of 0. The Raw score was the total of item score.
  Score range 0-29. Higher scores reflect better short term memory
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Test | Control
Number analyzed (Participants) | 185 | 178
Score on a scale | 2.86 (2.924) | 3.03 (2.813)

ADVERSE EVENTS:
Description: Safety population, defined as all participants who were randomized and administered at least one study treatment during the study. The population of analysis was safety population (N=524).
Arm/Group | Test | Control
Serious Adverse Events (participants affected / at risk) | 0/259 | 3/265
Other Adverse Events (participants affected / at risk) | 30/259 | 33/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test (N=259) | Control (N=265)
CONVULSION (Nervous system disorders) | 0 (0) | 1 (1)
STATUS EPILAPTICUS (Nervous system disorders) | 0 (0) | 1 (1)
ACUTE GASTRO ENTERITIS (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test (N=259) | Control (N=265)
NASOPHARYNGITIS (Infections and infestations) | 9 (9) | 10 (10)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 (7) | 10 (10)
PYODERMA (Infections and infestations) | 1 (1) | 0 (0)
VARICELLA (Infections and infestations) | 1 (1) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 3 (3)
IMPETIGO (Infections and infestations) | 0 (0) | 1 (1)
TYPHOID FEVER (Infections and infestations) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 6 (6) | 6 (6)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 3 (3)
NAUSEA (Infections and infestations) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 3 (3) | 8 (8)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.